CLINICAL TRIAL: NCT03549273
Title: Evaluation of the Effect of the Combination of the Natural Products Glizigen® and Ocoxin®-Viusid® in the Treatment of High-grade Cervical Intraepithelial Lesions. Phase II
Brief Title: Evaluation Glizigen® and Ocoxin®-Viusid® in High-grade Cervical Intraepithelial Lesions
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OOS-GLZ-2018
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma; Neoplasia; Intraepithelial, Cervix; Glandular Neoplasms; Epithelial Neoplasm; Neoplasms
Keywords: carcinoma; intraepithelial cervix lesions; Oxidative Stress; Ocoxin Viusid; Glizigen Spray
MeSH Terms: conditions — Carcinoma; Uterine Cervical Dysplasia; Neoplasms, Glandular and Epithelial; Neoplasms | interventions — Ocoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Glizigen® spray + Ocoxin-Visuid® oral solution
  Interventions: Dietary Supplement: Glizigen® + Ocoxin-Viusid®

INTERVENTIONS:
Dietary Supplement: Glizigen® + Ocoxin-Viusid® — * Glizigen® spray, topical use, 2 times a day for 6 months with an interruption for 2 months at the end of the third month.
  * Ocoxin®-Viusid® 60 ml daily (1 vial every 12 hours) by oral route for 8 months, preferably administered after breakfast and lunch, without interruption.

SUMMARY:
Phase II clinical trial, monocentric, not controlled, in patients with high grade cervical intraepithelial lesions. A total of 62 patients with a diagnosis of CIN II, III or carcinoma in situ will be included. It is expected that with the combination of natural products Glizigen® and Ocoxin®-Viusid® at least 60% of patients with treated intraepithelial lesions (IEL) have a global response (complete or partial), with elimination of the human papillomavirus and the viral load.

DETAILED DESCRIPTION:
Main objective: To evaluate the effect of the combination of Glizigen® and Ocoxin®-Viusid® in the treatment of high-grade cervical intraepithelial lesions. Specific objectives: 1. To evaluate the overall response (colposcopic, histological and virological) in patients treated with the combination of the natural products Glizigen® and Ocoxin®-Viusid® in the treatment of high-grade cervical intraepithelial lesions. 2. Evaluate the colposcopic response in patients treated with the combination of natural products. 3. Evaluate the histological response in patients treated with the combination of natural products after conization. 4. Evaluate the virological response in patients treated with the combination of natural products. 5.Describe adverse events during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that meet the diagnostic criteria.
2. Patients with age ≥18 years.
3. Patients with residual lesion greater than 3 mm after the initial punch, measurable by video colposcopy and with major changes (Criteria from Rio 2011).
4. Patients that have a positive test to the oncogenic virus of the human papilloma (16, 18, 31, 33, 45, 52 and 58).
5. Patients who give their informed consent to participation in writing.
6. Patients who consent to perform the conization according to the study schedule.
7. Patients with normal laboratory parameters within the limits established in the institution (complete blood count, platelets and erythrosedimentation. In the case of male sex (vasectomy, use of condoms) while the treatment lasts.

Exclusion Criteria:

1. Patients who have received surgical, ablative, radiant, immunomodulatory or chemotherapy treatment 30 days before recruitment.
2. Patients pregnant or breastfeeding.
3. Patients with acute cervico-vaginal infections.
4. Patients with positive serology known to HIV and/or syphilis.
5. Patients with diseases that compromise the state of consciousness or their possibility of collaboration.
6. Patients with a history of severe allergic history.
7. Patients who are participating in another research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Lesion progression | 9 months
  Colonoscopy. The categories will analyze as:
  * Complete Response-CR (Disappearance of the initial lesion and no new lesions appear).
  * Partial Response-PR (Reduction between 30 to 50% or more of the initial lesion and no new lesions appear).
  * Stable disease-SD (Same morphometry or reduction of less than 30% of the initial lesion).
  * Progressive Disease-PD (Increase in the diameter of the lesion The lesion extends to one or more quadrants that were not in the initial lesion. It will be considered progressive disease when at least two of the response variables are present.The variable viral load will always be present).
Lesion progression | 9 months
  Histology. The categories will analyze as:
  * CR (Disappearance of the initial lesion No degree of Cervical intraepithelial Neoplasia (CIN)).
  * PR (Reduction of CIN to one degree or more).
  * SD (Same degree of initial lesion is maintained).
  * PD (Increase in one degree of the lesion of CIN or presence of histological signs of invasion] It will be considered progressive disease when at least two of the response variables are present. The variable viral load will always be present).
Lesion progression | 9 months
  Virological. The categories will analyze as:
  * CR (Viral genotype- VG: Negative Human Papillomavirus (HPV) detection high or low oncogenic risk and Viral load: Not detectable).
  * PR (VG: No detection of viral genotypes of high oncogenic risk identified in the initial examination, but positive to HPV of low oncogenic risk Viral load: Reduction of the value of the viral load in at least one base logarithm 10).
  * SD (VG: Initial genotypes are maintained Viral load: Equal result than the initial examination, no change in the viral load values).
  * PD (VG: Initial genotypes or appearance of one or more oncogenic genotypes are maintained Viral load: Initial genotypes show an increase in viral load value in at least one base 10 logarithm. Other oncogenic genotypes appear with viral load values greater than or equal to 103 copies / ml.] It will be considered progressive disease when at least two of the response variables are present.The variable viral load will always be present).

SECONDARY OUTCOMES:
Colposcopy response | 9 months
  Complete Response: Disappearance of the initial lesion and no new lesions appear; Partial Response: Reduction between 30 to 50% or more of the initial lesion and no new lesions appear; Stable Disease: Equal morphometry or minor reduction 30% of the initial lesion; Progressive Disease: Increased diameter of the lesion The lesion extends to one or more quadrants that were not in the initial lesion).
Histological Response | 9 months
  Complete Response: Disappearance of initial injury No degree of CIN; Partial Response: Reduction of CIN to one degree or more; Stable Illness: Same degree of initial injury remains; Progressive Disease: Increase by one degree lesion of CIN or presence of histological signs of invasion).
Virological response | 9 months
  Complete response: Viral genotype: Negative result for the detection of human papillomavirus (HPV) with high or low oncogenic risk and Viral load: Not detectable; Partial response: Viral genotype: No detection of viral genotypes of high oncogenic risk (16, 18, 31 , 33, 45, 52 and 58) identified in the initial examination, but positive to HPV of low oncogenic risk and viral load: Reduction of the value of the viral load in at least one logarithm of base 10; Stable Disease: Viral genotype: Se maintain the initial genotypes and viral load: Same result as the initial examination, no change in the viral load values; Progressive Disease: Viral genotype: The initial genotypes are maintained or the appearance of one or more oncogenic genotypes and viral load: genotypes initials show an increase in the viral load value in at least one logarithm of base 10. Other oncogenic genotypes appear with viral load values greater than or equal to 103 copies/ml)
Adverse Events (AE) | 9 months
  The AE will measure as: -Occurrence of an AE in the patient (Yes/No) -Description of the AE (Name of the AE presented) -Duration of the AE (Difference of dates between the start and end of the AE) -Intensity of the AE (Classification according to CECMED Regulation 45/2007 in: Mild, Moderate, and Severe) -Gravity of AE (Serious or Not serious. Considering serious adverse events those that: 1.Produce the patient' death, 2.Life-threatening, 3.Hospitalization or prolongation of hospitalization indicated, 4. Produce significant or persistent disability, 5.Produce birth defect or congenital anomaly) -Attitude respect to the treatment under study (No changes, Dose modification, Temporary interruption of the treatments under study, Definitive interruption of the treatments under study). -Result of the EA (Recovered, improved, persists or sequels) -Causality Relationship (Definitive, Very likely, Probable, Possible, Not related, Unknown)

CONTACTS AND LOCATIONS:
Locations (1):
- Our Lady of Rule No. 52 &/Remedios and Quiroga, Luyano, Havana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] de Villiers EM. Cross-roads in the classification of papillomaviruses. Virology. 2013 Oct;445(1-2):2-10. doi: 10.1016/j.virol.2013.04.023. Epub 2013 May 16. PMID 23683837
- [Background] A'Hern RP. Sample size tables for exact single-stage phase II designs. Stat Med. 2001 Mar 30;20(6):859-66. doi: 10.1002/sim.721. PMID 11252008
- [Background] Bornstein J, Bentley J, Bosze P, Girardi F, Haefner H, Menton M, Perrotta M, Prendiville W, Russell P, Sideri M, Strander B, Tatti S, Torne A, Walker P. 2011 colposcopic terminology of the International Federation for Cervical Pathology and Colposcopy. Obstet Gynecol. 2012 Jul;120(1):166-72. doi: 10.1097/AOG.0b013e318254f90c. PMID 22914406
- [Background] Hernandez-Garcia S, Gonzalez V, Sanz E, Pandiella A. Effect of Oncoxin Oral Solution in HER2-Overexpressing Breast Cancer. Nutr Cancer. 2015;67(7):1159-69. doi: 10.1080/01635581.2015.1068819. Epub 2015 Aug 4. PMID 26241555
- [Background] Diaz-Rodriguez E, Hernandez-Garcia S, Sanz E, Pandiella A. Antitumoral effect of Ocoxin on acute myeloid leukemia. Oncotarget. 2016 Feb 2;7(5):6231-42. doi: 10.18632/oncotarget.6862. PMID 26756220
- [Background] Vilar Gomez E, Gra Oramas B, Soler E, Llanio Navarro R, Ruenes Domech C. Viusid, a nutritional supplement, in combination with interferon alpha-2b and ribavirin in patients with chronic hepatitis C. Liver Int. 2007 Mar;27(2):247-59. doi: 10.1111/j.1478-3231.2006.01411.x. PMID 17311621
- [Background] Stillo M, Carrillo Santisteve P, Lopalco PL. Safety of human papillomavirus vaccines: a review. Expert Opin Drug Saf. 2015 May;14(5):697-712. doi: 10.1517/14740338.2015.1013532. Epub 2015 Feb 18. PMID 25689872